CLINICAL TRIAL: NCT05405699
Title: 'Digitalization in Psychoeducation' The Effect of Tele-Psychoeducation on Problem-Solving Skills and Stress: A Randomized Factorial Trial
Brief Title: 'Digitalization in Psychoeducation' The Effect of Tele-Psychoeducation on Problem-Solving Skills and Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Gizem Beycan Ekitli, PhD., Research Assistant, Ege University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: EgeTrial2
Record Dates: First submitted 2022-06-01; First posted 2022-06-06 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Stress; Problems Psychosocial
Keywords: Problem solving skills; psychoeducation; stress; mobile health; telepsychiatry; digitalization

STUDY DESIGN:
Intervention Model Description: The study is a single-blind, randomized, factorial experimental type follow-up study with a control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Intervention (Experimental)
  Interventions: Behavioral: digitalized group psychoeducation

INTERVENTIONS:
Behavioral: digitalized group psychoeducation — Problem Solving Approach based problem solving skills psychoeducation's session topics of eight weeks are as follows:
  1. Introduction and warm-up,
  2. Problem orientation-identifying the problem,
  3. Identifying prior problems-Which do I want to start from?
  4. Recognizing the losses caused by problems and complaints,
  5. Setting reachable and realistic goals,
  6. Generating alternatives -What can I do?
  7. Regulating emotions,
  8. Experimenting and exploring. The main outcomes of each session were determined, and sessions were completed in approximately one hour as a semi-structured interactive group training according to group dynamics.
  Three days a week for eight weeks, informative posts were shared, asynchronous testing and self-discovery activities were carried out, and a synchronous tele-psychoeducation session was held once a week. Participants were connected to the live broadcast of the research team and interacted via text messages.
  Arms: Intervention

SUMMARY:
The effect of tele-psychoeducation based on an online social media platform, which had never been done previously, on problem-solving skills and stress levels in young adults was investigated. A randomized, single-blind factorial trial was conducted with two groups of 54 university students who met the inclusion criteria. Cognitive behavioural based psychoeducation was carried on via Instagram's both online and asynchronized sessions for 8 weeks. Data were collected using pre-/posttest and follow-up measurements with the Problem-Solving Inventory and Perceived Stress Scale and were analysed using factorial analysis of variance. ηp2 and Cohen's r was used, which shows the effect size with variance distribution.

DETAILED DESCRIPTION:
The research hypotheses are as follows:

1. H1: There is a significant difference between the mean scores of the Problem Solving Inventory in favour of the intervention group in the time series.
2. H1: There is a significant difference between the mean scores of the Perceived Stress Scale in favour of the intervention group in the time series.
3. H1: The recently developed group tele-psychoeducational intervention is effective for reducing Problem Solving Inventory mean scores.
4. H1: The recently developed group tele-psychoeducational intervention is effective for reducing Perceived Stress Scale mean scores.

Research data was collected with an online survey tool (Googledocs) that does not require a usage fee or license. The tool is convenient and economical in that it is suitable for use with any electronic device that can connect to the internet. The developed online form was piloted with ten students. Arrangements were made for the clarity of the questions and the convenience of the online tool. Pilot study data was not included in the findings. The tools detailed below were used to collect the data.

Personal Data Collection Form: This form consists of 11 multiple-choice questions to determine the variables that may have an impact on the sociodemographic characteristics, health history, and problem-solving skills of the participants. The questions were prepared by the research team in the light of the literature.

Problem Solving Inventory: The Problem Solving Inventory (PSI), developed by Heppner and Petersen (1982), is a Likert-type scale, scored between 1 and 6, consisting of 35 items that measure adults' self-perception of problem solving skills. There are items that are reverse coded and excluded from scoring. The higher total scores obtained from the scale indicate that the individual perceives himself as inadequate in terms of problem solving skills. The Cronbach alpha consistency coefficient of the original scale was .90, and the coefficients obtained for the subscales were between .72 and .85. The scale was adapted to Turkish by Şahin et al. (1993), and the Cronbach alpha consistency coefficient was found to be .88. In our study, the Cronbach alpha coefficient was .78.

Perceived Stress Scale: The scale was developed by Cohen et al. (1983), and adapted into Turkish by Eskin et al. (2013). The Perceived Stress Scale (PSS) is designed to measure how stressful situations in one's life are perceived. Five-point Likert-type scale items are interpreted over the total score and two sub-dimensions (Perception of Insufficient Self-efficacy and Perception of Stress Discomfort). A high total score indicates that the person perceives the stress he/she has been loaded with as high; it is interpreted as the methods used in coping with stress are not functional, and therefore they cannot cope with stress effectively. In our study, the Cronbach's alpha coefficient of the scale was determined as .75.

Data Collection: Data collection in the study was planned in line with the Checklist for Reporting Results of Internet E-Surveys (CHERRIES), which can be considered as a method and reporting guide for online survey research. The research's data security was ensured via a user account to which only two members of the research team had access and which would not be shared with any other user, and the access link was terminated when the data collection process was completed.

ELIGIBILITY:
Inclusion Criteria:

* Being adult
* Being volunteer to participation
* Must be have the required technological opportunities

Exclusion Criteria:

* To receive a professional support that can affect coping skills during the data collection process
* Not participate in 20% of tele-psychoeducational interventions

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Problem Solving Inventory (first evaluation with posttest) | Through study completion, an average of 4 months
  The Problem Solving Inventory (PSI), developed by Heppner and Petersen (1982), is a Likert-type scale, scored between 1 and 6, consisting of 35 items that measure adults' self-perception of problem solving skills. There are items that are reverse coded and excluded from scoring. The higher total scores obtained from the scale indicate that the individual perceives himself as inadequate in terms of problem solving skills. The Cronbach alpha consistency coefficient of the original scale was .90, and the coefficients obtained for the subscales were between .72 and .85 (Heppner & Petersen, 1982). The scale was adapted to Turkish by Şahin et al. (1993), and the Cronbach alpha consistency coefficient was found to be .88. In our study, the Cronbach alpha coefficient was .78.
Perceived Stress Scale (first evaluation with posttest) | Through study completion, an average of 4 months
  The scale was developed by Cohen et al. (1983), and adapted into Turkish by Eskin et al. (2013). The Perceived Stress Scale (PSS) is designed to measure how stressful situations in one's life are perceived. Five-point Likert-type scale items are interpreted over the total score and two sub-dimensions (Perception of Insufficient Self-efficacy and Perception of Stress Discomfort). A high total score indicates that the person perceives the stress he/she has been loaded with as high; it is interpreted as the methods used in coping with stress are not functional, and therefore they cannot cope with stress effectively. In our study, the Cronbach's alpha coefficient of the scale was determined as .75.
Problem Solving Inventory (second evaluation with follow up) | Through study completion, an average of 7 months
Perceived Stress Scale (second evaluation with follow up) | Through study completion, an average of 7 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University Faculty of Nursing, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes